CLINICAL TRIAL: NCT03623997
Title: Defining Systemic Control of Iron Absorption to Optimize Oral Iron Supplementation Regiemns for Women With Iron Deficiency Anemia
Brief Title: Measuring Erythrocyte Iron Incorporation From Different Dosing Regimens in Anemic Women
Status: Completed | Type: Observational
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof. Dr. med, Swiss Federal Institute of Technology
Other Study IDs: FeSupp_Anemia
Record Dates: First submitted 2017-11-06; First posted 2018-08-09 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Sulfates

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stable isotope labeled iron II sulfate: All subjects will go through two iron absorption study cycles. In one cycle they get 100mg oral iron labeled with stable isotopes on two consecutive and on one alternate day and in another cycle they get 200mg oral iron labeled with stable isotopes on two consecutive and on one alternate day. Half of the subjects start with the 100mg cycle whereas the other half starts with the 200mg cycle.
  Interventions: Other: Iron stable isotope labeled iron(II) sulfate

INTERVENTIONS:
Other: Iron stable isotope labeled iron(II) sulfate — Administration of oral stable isotope labels using different dosings and different regimens in women with iron deficiency anemia

SUMMARY:
Iron-deficient anaemic subjects are likely to benefit most from oral iron supplements, but supplementation schedules vary widely in clinical practice, absorption is low and compliance is poor due to mild gastrointestinal side effects. The investigators will compare iron absorption from labeled oral iron doses of 100mg and 200mg administered either on two consecutive days or on alternate days in young anemic women.

ELIGIBILITY:
Inclusion Criteria:

* Ferritin <15 µg/L
* Hb 8-11.9 g/dl
* BMI 18.5-24.9 kg/m2
* Body weight <70 kg

Exclusion Criteria:

* Severe anemia (Hb <8 g/dl)
* Elevated CRP >5.0 mg/L
* Chronic disease
* Long-term medication, except contraception
* Consumption of Mineral and Vitamin supplements within the study period
* Therapeutic iron infusion over the past 6 months
* Pregnancy or breastfeeding
* Smoking

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young women with iron-deficiency anemia
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Fractional and total iron absorption | absorption will be measured 14days after the 100mg and 200mg cycle
  Fractional and total iron absorption from different supplementation regimens
Serum hepcidin | right before the administration of an iron dose
  Serum hepcidin after the administration of different doses and using different regimens
Serum EPO | right before the administration of an iron dose
  Serum EPO after the administration of different doses and using different

SECONDARY OUTCOMES:
Serum ferritin | right before the administration of an iron dose
  Determination of iron status
Serum TfR | right before the administration of an iron dose
  Determination of iron status
Serum CRP | right before the administration of an iron dose
  Determination of inflammation status
Serum AGP | right before the administration of an iron dose
  Determination of inflammation status
Serum iron | right before the administration of an iron dose
  Determination of iron status
Total iron binding capacity | right before the administration of an iron dose
  Determination of iron status

CONTACTS AND LOCATIONS:
Locations (1):
- Human Nutrition Laboratory ETH Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Stoffel NU, Zeder C, Brittenham GM, Moretti D, Zimmermann MB. Iron absorption from supplements is greater with alternate day than with consecutive day dosing in iron-deficient anemic women. Haematologica. 2020 May;105(5):1232-1239. doi: 10.3324/haematol.2019.220830. Epub 2019 Aug 14. PMID 31413088